CLINICAL TRIAL: NCT02492646
Title: Effect of Normal Saline Lubrication of Endotracheal Tube on Post-intubation Complications: A Prospective Non-inferiority Trial
Brief Title: Effect of Saline Lubrication on Post-intubation Complications
Acronym: Lubrication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong-Hwa Seo, Pf., Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: JHSeo_Saline
Record Dates: First submitted 2015-07-01; First posted 2015-07-09 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2017-06

CONDITIONS: Postoperative Sore Throat

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Saline group (Experimental): In the saline group, disposable endotracheal tube was immersed in the 1 liter of sterile 0.9% sodium chloride irrigation solution before anesthetic induction.
  Interventions: Procedure: Saline group
- Dry group (Experimental): In the dry group, endotracheal tube was peeled off from sterile packing just before orotracheal intubation.
  Interventions: Procedure: Dry group

INTERVENTIONS:
Procedure: Saline group — After anesthetic induction, patients will be intubated with endotracheal tube which was immersed in normal saline before intubation.
  Arms: Saline group
Procedure: Dry group — After anesthetic induction, patients will be intubated with endotracheal tube which was not immersed in normal saline.
  Arms: Dry group

SUMMARY:
The purpose of this study is to evaluate the influence of none-lubricated dry tube on the incidence of Postoperative Sore Throat (POST) after general anesthesia with endotracheal intubation.

ELIGIBILITY:
Inclusion Criteria:

* patients aged between 20-80 years who were scheduled for surgery under general anesthesia requiring orotracheal intubation

Exclusion Criteria:

* history of gastroesophageal reflux disease (GERD)
* congenital or acquired abnormalities of the upper airway such as tumor, polyp, trauma, abscess, inflammation, infection, or foreign bodies
* previous airway surgery; increased risk of aspiration
* coagulation disorders
* previous history of difficult intubation or conditions with expected difficult airway including Mallampati classification ≥ 3 or thyromental distance < 6.5 cm
* Using the other intubation devices beyond the direct laryngoscopy such as lighted stylet or fiberoptic bronchoscopy
* symptoms of sore throat or upper respiratory tract infection
* expected to place nasogastric tube during perioperative period
* requiring nasotracheal intubation

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
incidence of postoperative sore throat (POST) | until one day after surgery
  ask patients whether they have sore throat after surgery

SECONDARY OUTCOMES:
Oropharyngeal injury | 2 hours and 24 hours after surgery
  assessed by direct visualization of the oropharyngeal cavity with regard to the location such as pharyngeal wall, uvula, vallecular, tonsillar fossa and pillars and presence of hyperemia, edema, hematoma, or any other lesions
respiratory symptoms | 1 week after the surgery
  At the 1 week postoperative follow-up phone call, patients would be asked if they have upper respiratory symptoms such as cough, sputum, sore throat or fever. And if so, they would be checked if they diagnosed following diseases, common cold, tonsillitis, pneumonia or any other possible respiratory infectious diseases.
severity of postoperative sore throat (POST) | When arriving at postanesthesia care unit (PACU) and thereafter 2, 4, and 24 hours after the surgery
  The severity of POST was evaluated on a 4-point-scale : 0, no sore throat; 1, mild sore throat (complained of sore throat only upon inquiry); 2, moderate sore throat (complained of sore throat on his/her own); 3, severe sore throat (change of voice or hoarseness, associated with throat pain)

CONTACTS AND LOCATIONS:
Overall Officials: Jeong-Hwa Seo, Associate professor, Study Chair — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim E, Yang SM, Yoon SJ, Bahk JH, Seo JH. The effects of water lubrication of tracheal tubes on post-intubation airway complications: study protocol for a randomized controlled trial. Trials. 2016 Nov 25;17(1):562. doi: 10.1186/s13063-016-1699-0. PMID 27887662